CLINICAL TRIAL: NCT00815958
Title: Embolic Events Detected During Total Knee Arthroplasty With and Without the Use of RIA (Reamer-Irrigator-Aspirator): A Blinded, Randomized, Controlled Clinical Study
Brief Title: Embolic Events Detected During Total Knee Arthroplasty With the Use of RIA (Reamer-Irrigator-Aspirator)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: administrative reasons
Sponsor: Ohio State University (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2007H0111; 60013485
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Total Knee Replacement
Keywords: knee replacement surgery; Reamer-Irrigator-Aspirator; femoral reaming; fat embolism
MeSH Terms: conditions — Embolism, Fat

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Reaming with Synthes RIA (Reamer-Irrigator-Aspirator)
  Interventions: Procedure: Reaming with Synthes RIA (Reamer-Irrigator-Aspirator)
- B (Active Comparator): Reaming with conventional reamer
  Interventions: Procedure: Reaming with conventional reamer

INTERVENTIONS:
Procedure: Reaming with Synthes RIA (Reamer-Irrigator-Aspirator) — During knee replacement surgery, the study anesthesiologist will place probes for the transesophageal echocardiogram (TEE) and the transcranial Doppler ultrasound (TCD). In patients randomized to the RIA group (Arm A), surgery performed by the investigating orthopaedic surgeon will be done according to standard of care guidelines up until femoral reaming. These patients will receive reaming with RIA. The remainder of the surgery will also be done according to the standard of care. TEE and TCD data will be recorded throughout the surgery.
  Other Names: Synthes Reamer-Irrigator-Aspirator; RIA
  Arms: A
Procedure: Reaming with conventional reamer — During knee replacement surgery, the study anesthesiologist will place probes for the transesophageal echocardiogram (TEE) and the transcranial Doppler ultrasound (TCD). In patients randomized to the control group (Arm B), surgery performed by the investigating orthopaedic surgeon will be done according to standard of care guidelines. These patients will receive reaming with the conventional method/reamer. TEE and TCD data will be recorded throughout the surgery.
  Other Names: Synthes Reamer-Irrigator-Aspirator; RIA
  Arms: B

SUMMARY:
The embolisation of fat and bone marrow during long bone instrumentation is a well-known complication of major joint replacement surgery. Clinically significant venous thromboembolic disease, cardiopulmonary dysfunction,cerebral emboli, and death have all been described. Because the intravasation of medullary contents is caused by increased pressure during canal instrumentation, the use of the Synthes RIA (Reamer-Irrigator-Aspirator), a negative pressure-irrigated high-speed reamer, may result in a lower incidence of embolism.

This controlled clinical trial will evaluate the utility of the RIA in reducing the frequency and severity of embolic events as detected by intraoperative transesophageal echocardiography (TEE) and transcranial Doppler (TCD) during total knee arthroplasty (TKA) surgery.

DETAILED DESCRIPTION:
Patients scheduled to undergo total knee replacement surgery will be randomized to receive reaming with either the Synthes RIA (intervention group) or standard reamer (control group). All subjects will undergo intraoperative monitoring with transesophageal echocardiography and transcranial Doppler ultrasound. Both intraoperative and postoperative oxygen saturation levels will be monitored and recorded for evidence of hypoxemia. Subjects will be evaluated for evidence of thrombogenesis and systemic inflammation both preoperatively and at selected postoperative intervals.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Scheduled or soon to be scheduled for elective total knee replacement surgery
* No previous history of hip or (ipsilateral) knee replacement

Exclusion Criteria:

* Subject is under 18
* Prior instrumentation of the medullary canal (knee or hip)
* History of esophageal or GI disease or other contraindication for TEE
* Previous history of DVT
* Currently on anti-coagulant therapy (i.e. Coumadin or others)
* Currently on supplemental oxygen or SpO2 is below 90 on room air
* Cognitive or language barriers limiting comprehension of study materials in English
* Subject is pregnant or planning pregnancy
* Current or impending incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The incidence of intraoperative embolic events detected with transesophageal echocardiography and transcranial Doppler and the grade or size of these embolic events | During surgery

SECONDARY OUTCOMES:
Activation of thrombogenesis and VTE complications, intraoperative and postoperative hypoxemia, and level of systemic inflammation. | Post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cornel Van Gorp, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, University Hospital East, Columbus, Ohio, United States